CLINICAL TRIAL: NCT02928341
Title: Impact Evaluation of Urban Water Supply Improvements on Cholera and Other Diarrhoeal in Uvira, Democratic Republic of Congo
Brief Title: Impact Evaluation of Urban Water Supply Improvements on Cholera and Other Diarrhoeal Diseases in Uvira, Democratic Republic of Congo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 8913
Record Dates: First submitted 2016-10-07; First posted 2016-10-10 (Estimated); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Cholera; Diarrhea
MeSH Terms: conditions — Cholera; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No intervention (No Intervention): Current water supply access
- Intervention (Experimental): Received water supply improvement intervention designed to improve access to tap water, consisting of community managed public taps, improved tap water distribution network, refurbished tap connections and promotion of new household tap connections.
  Interventions: Other: Improved water supply

INTERVENTIONS:
Other: Improved water supply
  Arms: Intervention

SUMMARY:
The aim of the study is to evaluate the impact of a large-scale urban water supply improvement intervention on cholera and other diarrhoeal diseases. The study uses a step wedge cluster randomised controlled trial (SWcRCT) to measure the effect of the intervention on cholera centre admission rates and confirmed cholera cases. A nested cohort study will examine changes in water-related practices following the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Uvira resident admitted to the Uvira Cholera Treatment Centre in Uvira

Exclusion Criteria:

* Any patients admitted during the period of intervention implementation in each cluster

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4556 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Admission rate to the Uvira Cholera Treatment Centre | 36 months

SECONDARY OUTCOMES:
Admission rate to the Uvira Cholera Treatment Centre of laboratory confirmed cholera cases | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Cumming, MSc, Principal Investigator — London School of Hygiene and Tropical Medicine; Karin Gallandat, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Centre de Traitement du Cholera, Hôpital General de Reference d'Uvira, Sud-Kivu, République Démocratique du Congo, Uvira, South Kivu, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gallandat K, Macdougall A, Jeandron A, Mufitini Saidi J, Bashige Rumedeka B, Malembaka EB, Azman AS, Bompangue D, Cousens S, Allen E, Cumming O. Improved water supply infrastructure to reduce acute diarrhoeal diseases and cholera in Uvira, Democratic Republic of the Congo: Results and lessons learned from a pragmatic trial. PLoS Negl Trop Dis. 2024 Jul 3;18(7):e0012265. doi: 10.1371/journal.pntd.0012265. eCollection 2024 Jul. PMID 38959264
- [Derived] Gallandat K, Jeandron A, Ross I, Mufitini Saidi J, Bashige Rumedeka B, Lumami Kapepula V, Cousens S, Allen E, MacDougall A, Cumming O. The impact of improved water supply on cholera and diarrhoeal diseases in Uvira, Democratic Republic of the Congo: a protocol for a pragmatic stepped-wedge cluster randomised trial and economic evaluation. Trials. 2021 Jun 21;22(1):408. doi: 10.1186/s13063-021-05249-x. PMID 34154636
- [Derived] Williams C, Cumming O, Grignard L, Rumedeka BB, Saidi JM, Grint D, Drakeley C, Jeandron A. Prevalence and diversity of enteric pathogens among cholera treatment centre patients with acute diarrhea in Uvira, Democratic Republic of Congo. BMC Infect Dis. 2020 Oct 9;20(1):741. doi: 10.1186/s12879-020-05454-0. PMID 33036564